CLINICAL TRIAL: NCT07224217
Title: Evaluating a Remotely Delivered Physical Activity Program for Inactive Men in Rural Communities: A Feasibility Study
Brief Title: Remote Exercise Program for Rural Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000136
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rural Health
Keywords: physical activity; behavioral intervention; Rural men
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Receive intervention immediately after randomization
  Interventions: Behavioral: Remote Physical Activity Program (12 weeks)
- Delayed (Other): Start intervention after 12 week assessment
  Interventions: Behavioral: Delayed Remote Physical Activity Program (6 weeks)

INTERVENTIONS:
Behavioral: Remote Physical Activity Program (12 weeks) — Participants will receive a 12 week remotely delivered physical activity program immediately after randomization. Participants will receive bi-weekly calls, behavioral lessons, and bi-weekly behavioral feedback via email.
  Arms: Immediate
Behavioral: Delayed Remote Physical Activity Program (6 weeks) — Participants receive a 6 week remote physical activity program after completing the 12 week assessment. The program includes weekly calls, behavioral lessons, and weekly behavioral feedback via email.
  Arms: Delayed

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of a remote physical activity intervention designed for rural inactive men.

DETAILED DESCRIPTION:
The proposed study is a pilot randomized controlled trial that will randomize participants to either 1) Immediate intervention, which consists of a 12-week physical activity program or 2) Delayed Intervention, which participants will be assigned to a 6-week abridged version of the program at the end of 12 weeks. Both versions of the physical activity program will provide participants a platform to report their exercise weekly, behavioral lessons, and receive personalized feedback on activity levels. The primary endpoint is to examine the feasibility and acceptability of the 12-week program by evaluating recruitment and retention rates, completion of phone calls, adherence to physical activity self-monitoring, and program satisfaction at 12-weeks. Preliminary efficacy will be assessed by changes in moderate-vigorous physical activity (MVPA), steps/day, health-related quality of life, self-efficacy, self-regulation, and supportive accountability at the end of 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Identify biological sex as male
* Engage in less than 90 minutes of self-reported moderate intensity exercise
* Ability to read and write in English
* Primarily living in a rural jurisdiction defined by 1 of the 7 more widely used definitions of rurality by the United States government
* Ability to walk independently for at least one block

Exclusion Criteria:

* Have a medical condition that could be made worse with a change in physical activity
* Plans to relocate from primary residence within 3 months of signing up for study
* Not willing to wear physical activity monitor for 7 days or complete surveys
* Less than 4 valid days of activity monitor wear time at baseline assessment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 12 weeks
  Percentage of recruitment rate (screened/enrolled)
Retention | 12 weeks
  Percentage of participants who complete the study
Adherence to coaching calls | 12 weeks
  Percentage of coaching calls completed in Immediate condition
Adherence to self-monitoring | 12 weeks
  Percentage of self-monitoring logs submitted in Immediate condition
Acceptability | 12 weeks
  Program satisfaction with the 12 week remote program in Immediate condition

SECONDARY OUTCOMES:
Physical activity - Moderate to vigorous minutes/week | baseline to 12 weeks
  Moderate-vigorous intensity physical activity (minutes/week) assessed by activPAL
Physical activity - Steps | baseline to 12 weeks
  Steps/day assessed by activPAL
Global Health | baseline to 12 weeks
  Global Health assessed via PROMIS (t-score)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Pellegrini, PhD, Study Director — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on request to the PI
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available on request after outcomes have been published
Access Criteria: IPD will be available on request after outcomes have been published